CLINICAL TRIAL: NCT01526863
Title: Assessment of the Effect of an HA Egg Administration for 6 Months on the Tolerance Induction to Egg in Children Allergic to Egg as Compared to a Placebo
Brief Title: Hydrolyzed Egg and Tolerance Induction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10.53.NRC
Record Dates: First submitted 2012-01-30; First posted 2012-02-06 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Allergy
Keywords: Allergy; Egg
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: HA egg
- HA egg (Active Comparator)
  Interventions: Dietary Supplement: HA egg

INTERVENTIONS:
Dietary Supplement: HA egg — Daily dose of HA egg or placebo for 6 months

SUMMARY:
The aim of this trial is to assess the effect of hydrolyzed egg orally administered on oral tolerance induction to egg in children allergic to egg as compared to a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Child of any ethnicity aged between 12 and 66 months at the time of enrolment

  * Positive Skin Prick Test (SPT) to egg white within the last 3 months
  * Either positive oral challenge OR convincing history, defined as an immediate (<1h) reaction following isolated ingestion of egg, positive SPT to egg white and positive sIgE (> 0.35 kU/L) for at least one of the following: egg, egg white, ovalbumin, ovomucoid, within the last 12 months
  * Having obtained his/her signed legal representative's informed consent.

Exclusion Criteria:

* History of severe anaphylaxis to egg

  * Significant pre-natal and/or post-natal disease
  * Child on systemic drugs (e.g. antihistamines, beta-agonists, ACE-inhibitors) according to half-life at time of enrolment
  * Congenital illness or malformation that may affect normal growth (especially immunodeficiency)
  * Child whose parents / caregivers cannot be expected to comply with treatment
  * Child currently participating in another interventional clinical trial

Ages: 12 Months to 66 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2012-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
positive or negative result (objective and subjective symptoms) of a challenge test with egg | 6 months

SECONDARY OUTCOMES:
compliance (product taken) | 6 months
skin prick test (sensitization to egg; size of wheal and flare) | 6 months
Immunological parameters: total and specific IgE and IgG4, cytokines, basophil activation | 6 months
Morbidity / Adverse Events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Papadopoulos, Prof., Study Chair — University of Athens, Greece; Antonella Muraro, Prof, Principal Investigator — University Hospital of Padua, Italy; Roger Lauener, Prof., Principal Investigator — Hochgebirgsklinik Davos, Switzerland; Stavroula Giavi, Dr., Principal Investigator — University of Athens, Greece
Locations (3):
- University of Athens, Athens, Greece
- University Hospital of Padua, Padua, Italy
- Hochgebirgsklinik Davos, Wolfgang, Switzerland